CLINICAL TRIAL: NCT01964859
Title: Feasibility Study for Fibroblast Autologous Skin Grafts: Biopsy of Skin Fibroblasts, Expansion in Cell Therapy Core, Topical Injection of Fibroblasts, and Subsequent Removal of Graft for Laboratory Studies.
Brief Title: Feasibility Study for Fibroblast Autologous Skin Grafts
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); United States Department of Defense (U.S. Federal Agency); Maryland Stem Cell Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00068684; 1R01AR064297-01A1 (NIH)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Wounds and Injuries
Keywords: healthy skin; wounds and injuries; prosthetics; amputations; dermal fibroblasts
MeSH Terms: conditions — Wounds and Injuries | interventions — ArteFill

STUDY DESIGN:
Masking Description: Sites are labeled as A, B and C and masked for outcomes assessors-- but these are all in the same subject.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous skin fibroblasts (Experimental): The investigators are comparing 3 injection sites in the same individual
  Interventions: Biological: autologous skin fibroblasts; Biological: Filler Product

INTERVENTIONS:
Biological: autologous skin fibroblasts — autologous skin fibroblasts
Biological: Filler Product — In some select subjects the investigators will test if the addition of an FDA approved filler product Bellafill might enhance cellular efficacy.
  Other Names: Bellafill

SUMMARY:
This research is being done to determine if investigators can change skin from one type to another. Specifically, investigators are interested in making normal skin into the thicker skin found on our palms and soles.

DETAILED DESCRIPTION:
To change the skin identity investigators propose to take skin cells from a person's own sole or palm (these are called "autologous skin fibroblasts"), multiply them in the lab, inject the cells (now called a "graft") back into the same person but at a different site of skin like the buttock, and then eventually remove the injected cells to see if they caused the skin to change.

Investigators hope that information from this study will help with problems like skin break-down in patients with amputations and prosthetics. The skin at their stump was not meant to withstand the pressure and friction of prosthetics and this study is the first step in trying to convert stump skin to palm/sole-like skin. In some select subjects the investigators will test if the addition of an FDA approved filler product might enhance cellular efficacy.

ELIGIBILITY:
Inclusion Criteria:

* May be male or female
* Must be between 18 years and 65 years of age
* In the opinion of the investigator, must be medically able to undergo the administration of study material determined by laboratory tests obtained within 7 days before baseline for which the investigator identified no clinically significant abnormality.
* Be able to comprehend the informed consent document and provide consent for participation
* Females of childbearing potential must:

  * have a negative pregnancy test at screening
  * agree to not become pregnant or breastfeed for the period of the study through 1 month after completion of the study
  * be willing to use a reliable form of contraception during the study
* Have healthy skin as determined by the PI or study Nurse Practitioner.
* Be willing and able to comply with the scheduled visits, biopsy/injection procedures, wound care instructions treatment plan, and other study procedures for the duration of the study.

Exclusion Criteria:

* Having received any investigational drug within 30 days prior to study entry
* An allergy history to any study materials including local anesthetic, dimethyl sulfoxide, human albumin, or bovine constituents, or hetastarch
* Pregnant, lactating, or trying to become pregnant
* A history of keloid formation
* An active nonhealing wound
* Having a significant medical history that the investigator feels is not safe for study participation (for example, some forms of autoimmune conditions, metastatic cancer, infectious diseases such as HIV, Human T-lymphotropic virus (HTLV) I/II, Hepatitis B, Hepatitis C). Biopsies taken from individuals with infections that are not allowed to enter the cell therapy core will make it such that these individuals cannot participate.
* Specifically we will exclude those with autoimmune diseases affecting the skin such as lupus.
* Having current skin diseases (i.e. extreme and active eczema, psoriasis, lichen planus) that the investigator feels is not safe for study participation
* A diagnosis of uncontrolled diabetes
* Active smoker during the study
* We will also exclude those who are on chronic immunosuppressive therapies such as oral steroids, but also those on chronic topical steroids in the area of investigation.
* Known bovine or meat sensitivity or severe allergies manifested by anaphylaxis to any product
* Known bleeding disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01-07 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Cytoplasmic size increase | 6 months
  Volar keratinocytes have larger area of the cytoplasm. We will quantitate the area of cytoplasm of non-volar keratinocytes to see if they increase selectively with volar fibroblasts as opposed to other fibroblasts injections or vehicle. The change in the area of cytoplasm of non-volar keratinocytes will be measured. The units of this measurement are a ratio of cytoplasmic area to total cellular area as a control.

SECONDARY OUTCOMES:
Durometer reading | 6 months
  Durometers measure the firmness of the skin. We will measure all sites to see if the area injected with volar fibroblasts is more firm. The units of measurement is in Durometer Units.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garza, MD, PhD, Principal Investigator — Department of Dermatology, Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Dermatology Department, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the requirements of the journal in which we finally publish.